CLINICAL TRIAL: NCT04839900
Title: A Cluster Randomized Controlled Trial of Pro-active Community Case Management for Malaria in Chadiza District, Eastern Province, Zambia
Brief Title: Proactive Community Case Management for Malaria in Zambia
Acronym: ProACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Ministry of Health, Zambia (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1704068
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Malaria, Falciparum; Malaria
Keywords: Malaria; integrated community case management; proactive response; Zambia
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: A two arm, cluster-randomized controlled trial (CRCT) will be conducted to determine whether proactive iCCM (arm 1)-- year-round weekly household visits by CHWs to test people of all ages with fever or history of fever with RDTs and offer treatment with an ACT for those who test positive (and treatment or referral of diarrhea and pneumonia for children under 5 years) -- compared to standard passive iCCM (arm 2)- malaria case management for all ages, and treatment or referral of diarrhea and pneumonia for children under 5 years, conducted by CHWs -- is associated with a greater reduction in confirmed malaria cases and parasite prevalence over a 2-year follow-up period. ]
  Clusters defined by CHW location will be randomly allocated to receive either proactive iCCM or standard passive iCCM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive iCCM (Active Comparator): Community health workers (CHWs) will conduct weekly visits of all households in their communities to detect children < 5 years with diarrhea or cough, and people of all ages complaining of fever or history of fever. Weekly household visits will be conducted year round. CHWs will be available for consultation throughout the week for sick visit consultations as per national iCCM policy (with malaria case management for all ages).
  Interventions: Other: Proactive iCCM
- Standard Passive iCCM (No Intervention): Community health workers (CHWs) will provide case management per national iCCM policy to all who are brought for consultation, but will not conduct household visits to provide active case detection. CHWs will be available for consultation throughout the week for sick visit consultations as per national iCCM policy (with malaria case management for all ages).

INTERVENTIONS:
Other: Proactive iCCM — CHWs in the proactive iCCM intervention arm will conduct weekly visits of all households in their communities to detect children < 5 years with diarrhea or cough, and people of all ages complaining of fever or history of fever. People with fever or history of fever in the past 48 hours, or any person with symptoms suggestive of malaria (chills, headache, muscle ache, fatigue, etc), will receive an RDT; those with positive results will be defined as confirmed malaria cases, and will receive the first line antimalarial. Any child under 5 years with diarrhea will be treated with oral rehydration solution (ORS) and zinc, and any child meeting diagnostic criteria for pneumonia will receive the first line antibiotic recommended per national iCCM policy. If the CHW does not have the indicated therapy on hand, the patient will be referred for treatment.
  Arms: Proactive iCCM

SUMMARY:
To study if a proactive strategy of weekly household visits by community health workers (CHWs) to identify people with malaria symptoms, offer diagnostic testing, and treatment for those with positive tests in Chadiza District, Eastern Province, can decrease malaria incidence and prevalence compared to conventional community case management.

DETAILED DESCRIPTION:
This study will be a two arm, cluster-randomized controlled trial to determine whether year round weekly household visits by CHWs to detect and test people of all ages with fever or history of fever with RDTs (and offer diagnosis and referral or treatment of diarrhea and pneumonia for children under 5 years), and offer treatment with an ACT for those who test positive compared to standard passive iCCM by CHWs (which includes malaria case management for all ages in Zambia), is associated with a greater reduction in confirmed malaria cases and parasite prevalence over a 2-year follow-up period.

Randomization will occur at the level of the CHW catchment areas. Thirty-three clusters will be enrolled in each arm for a total of 66 clusters. Primary study outcomes will be evaluated based on household-level cross-sectional surveys conducted at baseline and end-line and confirmed malaria case data collected through the health system throughout the study period.

Primary objectives:

1. Assess whether year-round weekly proactive iCCM compared to passive iCCM with malaria case management for all ages reduces the prevalence of patent (by rapid diagnostic test (RDT)) and subpatent (by PCR) parasitemia detected at the household level in cross sectional household surveys.
2. Determine whether the confirmed malaria case incidence (detected by CHWs (either proactively or passively) and at health facilities) decreases over time in communities with weekly proactive iCCM compared to passive iCCM by comparing the difference in slope of confirmed malaria incidence in proactive vs routine arms using an interrupted time series analysis

Secondary objectives:

1. Assess whether access to care (proportion of the population with fever in the past two weeks who received care from a qualified health provider, including community health worker), promptness of care (within 24 and 48 hours of symptoms), access to diagnostic malaria testing (proportion of the population with fever in the past two weeks who received a diagnostic test for malaria), and treatment with artemisinin-based combination therapy (ACT) if RDT is reported positive, is improved by proactive iCCM compared to passive iCCM
2. Describe the incidence of febrile disease, by arm, as well as the incidence of symptomatic malaria infection (febrile persons with a positive RDT), detected during proactive iCCM visits
3. Compare the incidence of malaria, by arm, detected at health facilities
4. Compare the proportion of malaria cases detected at community vs health facility, by arm
5. Determine if proactive iCCM reduces severe disease (malaria in all ages, diarrhea and pneumonia among < 5) compared to passive iCCM identified at health facility and community level)
6. Compare level of parasite exposure in intervention and control arms using multiplex bead based assay for long, medium and short duration antibodies
7. Determine programmatic cost per additional case detected and treated at the community level with proactive iCCM
8. Describe the feasibility, challenges, and benefits of proactive iCCM from the perspective of the facility health worker, CHW, and community members
9. Describe the benefits and challenges associated with incorporating diagnosis and treatment of pneumonia and diarrhea for children under 5 years

ELIGIBILITY:
All residents of all ages in the study area will be eligible to receive the CHW intervention.

All ages with fever

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10890 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Parasite Prevalence | 24 months
  1) Difference in parasite prevalence in intervention vs control clusters over time measured by RDT and PCR among all age groups (stratified by < 15 and 15+ years), detected through baseline and endline cross-sectional surveys conducted at the end of the transmission season.
Confirmed malaria case incidence | 24 months
  2) Difference in slope of trend lines of total numbers of febrile patients detected and malaria cases diagnosed monthly (CHWs + HF) in intervention vs control clusters (CHWs + HF)

CONTACTS AND LOCATIONS:
Locations (1):
- Chadiza District Health Office, Chadiza, Eastern Provice, Zambia

IPD SHARING:
Plan to Share IPD: Undecided
Future analyses might be required and an approval will be sought and granted by the local governing research ethics, Eres Converge, before such analyses can be performed. Any request for potential future secondary use will need review and approval by an IRB committee with full disclosure of the previous study protocol and Eres Converge committee reviews. Any transfer of samples and data to a collaborator or other agent/institute will be governed by the local rules and regulations, including those set forth by the Zambia National Health Research Authority for Material Transfer Agreements and the Ministry of Health in accordance with the Eres Converge.

REFERENCES:
- [Derived] Rutagwera MI, Ferriss EL, Kabamba BM, Porter T, Kangale CC, Gallalee S, Simataa M, Miller JM, Phiri-Chibawe C, Musunse M, Nyendwa P, Kapenda V, Psychas P, Gutman JR, Hawela M, Banda I, Chitambala-Otiono S, Bennett A, Hamainza B, Thwing JI. Impact of proactive malaria community case management (proCCM) on parasite prevalence and incidence from 2021 to 2023: a randomised controlled trial in Chadiza District, Eastern Province, Zambia. BMJ Glob Health. 2025 May 24;10(5):e017697. doi: 10.1136/bmjgh-2024-017697. PMID 40412814